CLINICAL TRIAL: NCT05768282
Title: Administration of Oral Prednisolone to Prevent Esophageal Stricture After Balloon-type Radiofrequency Ablation for Long-segment Esophageal Neoplasia
Brief Title: Oral Prednisolone to Prevent Esophageal Stricture After RFA for Long-segment Esophageal Neoplasia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EDAHS111018
Record Dates: First submitted 2022-10-10; First posted 2023-03-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Neoplasms; Esophagus Stenosis
Keywords: Esophageal stenosis; Esophageal squamous cell neoplasia; Endoscopic radiofrequency ablation; Prednisolone
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Stenosis | interventions — Prednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of oral prednisolone (Experimental): Oral prednisolone start at a dose of 30 mg/day on the third day after RFA, and continue for 4 weeks.
  Interventions: Drug: Oral prednisolone (30mg/day) for 28 days

INTERVENTIONS:
Drug: Oral prednisolone (30mg/day) for 28 days — Oral prednisolone was started at a dose of 30 mg/day on the third day after RFA, and continued for 4 weeks.
  Other Names: steroid

SUMMARY:
Endoscopic radiofrequency ablation (RFA) has shown good efficacy and safety in eradicating flat-type early esophageal squamous cell neoplasia (ESCN). However, post-RFA stricture is still a major concern, especially when treating long-segment early ESCNs. The aim of this study was to investigate the efficacy and safety of oral prednisolone to prevent post-RFA stricture.

DETAILED DESCRIPTION:
Esophageal cancer is the eighth most common cancer and the sixth most common cause of cancer death worldwide. The incidence rates of esophageal squamous cancers are still increasing in some countries in the Asia-Pacific region and Africa. Recently, image-enhanced endoscopy techniques such as Lugol or virtual chromoendoscopy have been shown to improve the detection and diagnosis of early esophageal squamous cell neoplasia (ESCN). However, some ESCNs spread laterally and present as long-segment lesions or appear with a mosaic pattern, all of which increase the difficulties and adverse event rates if treated by endoscopic resection. In particular, for extensive ESCNs, endoscopic submucosal dissection (ESD) has been associated with severe refractory stricture, even after pre-emptive steroid administration. This then requires repeated sessions of balloon dilation, leading to a decreased quality of life and increased medical expenses.

Radiofrequency ablation (RFA) has rapidly evolved in recent decades, and previous studies have shown its efficacy and safety in treating early ESCNs. Current evidence has shown that RFA is indicated for totally flat-type precancerous lesions, such as high-grade intraepithelial neoplasia (HGIN) or moderate-grade intraepithelial neoplasia (MGIN), or those that are not feasible for ESD. RFA is less technically demanding and more feasible for widely extended lesions. However, post-RFA esophageal stricture is still a concern, with an average frequency of 14~28%. The longitudinal length of the treatment area is the key factor associated with post-operative stricture. Around 50% of cases where the lesion is extended by more than 9 cm will develop post-RFA esophageal stricture, and thus a preventive strategy is urgently needed. The investigators previously evaluated the in vivo tissue effect of RFA by endoscopic ultrasound, and the results showed that the mucosa and submucosal layer were more edematous and thicker after RFA than before the procedure, suggesting that the thermal effect of RFA may injure the submucosa resulting in inflammation-related fibrosis and stricture. Steroids have an anti-inflammatory effect, and previous studies have shown that steroid treatment could potentially reduce post-ESD stricture in lesions occupying more than three-quarters of the circumference. However, the effectiveness of steroid treatment in preventing post-RFA stricture has yet to be elucidated. Therefore, the aim of this study is to investigate the effectiveness and safety of oral prednisolone treatment in preventing post-RFA esophageal stricture in long-segment and extensive ESCNs.

ELIGIBILITY:
Inclusion Criteria:

* Histology from endoscopic biopsies showed squamous intraepithelial neoplasia without stromal invasion;
* No lymph node metastasis on endoscopic ultrasound or computed tomography;
* Magnifying endoscopy showed the intraepithelial papillary capillary loop as type B1 pattern, according to the classification of the microvascular architecture of superficial esophageal carcinoma.

Exclusion Criteria:

* A prior history of endoscopic resection, radiation therapy or esophagectomy for esophageal cancer;
* A stricture that prevented the passage of a therapeutic endoscope;
* Uncontrolled coagulopathy;
* Poorly controlled diabetes mellitus.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with esophageal stenosis after RFA | at 1 month after the RFA procedure
  Defined as the failure of a standard endoscope (9.8 mm in diameter) to pass through the stenosis.Then the outcome measures will be compared with a historical control, that just received endoscopic surveillance.

SECONDARY OUTCOMES:
The number of endoscopic balloon dilatation sessions required | at 1 month after the RFA procedure
  f the esophageal stenosis was confirmed by endoscopy, balloon dilation will be done to resolve the symptoms
The adverse events rate | up to 1 year
  After oral prednisolone, the adverse events will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- EDA Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ono S, Fujishiro M, Niimi K, Goto O, Kodashima S, Yamamichi N, Omata M. Predictors of postoperative stricture after esophageal endoscopic submucosal dissection for superficial squamous cell neoplasms. Endoscopy. 2009 Aug;41(8):661-5. doi: 10.1055/s-0029-1214867. Epub 2009 Jun 29. PMID 19565442
- [Background] Yamaguchi N, Isomoto H, Nakayama T, Hayashi T, Nishiyama H, Ohnita K, Takeshima F, Shikuwa S, Kohno S, Nakao K. Usefulness of oral prednisolone in the treatment of esophageal stricture after endoscopic submucosal dissection for superficial esophageal squamous cell carcinoma. Gastrointest Endosc. 2011 Jun;73(6):1115-21. doi: 10.1016/j.gie.2011.02.005. Epub 2011 Apr 14. PMID 21492854
- [Background] Wang WL, Chang IW, Chen CC, Chang CY, Tseng CH, Tai CM, Lin JT, Wang HP, Lee CT. Lessons from pathological analysis of recurrent early esophageal squamous cell neoplasia after complete endoscopic radiofrequency ablation. Endoscopy. 2018 Aug;50(8):743-750. doi: 10.1055/s-0044-101352. Epub 2018 Feb 15. PMID 29448289
- [Background] Wang WL, Chang IW, Chen CC, Chang WL, Chu YY, Wu PH, Tai WC, Chen PY, Hsieh PH, Chung CS, Chang CY, Lin JT, Wang HP, Lee CT. Predictors for postoperative esophageal stricture after balloon-based radiofrequency ablation for early esophageal squamous neoplasia: a multicenter validation study. Therap Adv Gastroenterol. 2016 May;9(3):257-64. doi: 10.1177/1756283X16633051. Epub 2016 Feb 25. PMID 27134656
- [Derived] Wang WL, Tsai YN, Hsu MH, Lin JT, Wang HP, Lee CT. Administration of oral prednisolone to prevent esophageal stricture after balloon-type radiofrequency ablation for ultralong-segment esophageal neoplasia. Gastrointest Endosc. 2024 Aug;100(2):192-199. doi: 10.1016/j.gie.2024.03.030. Epub 2024 Apr 5. PMID 38583540